CLINICAL TRIAL: NCT03195998
Title: Determining the Validity of Transcutaneous Bilirubin Monitoring in Preterm Infants With a Gestational Age of 23 0/7 - 34 6/7 Weeks
Brief Title: Validity of Transcutaneous Bilirubin Monitoring in Preterm Infants
Acronym: TcB
Status: Completed | Type: Observational
Sponsor: Pediatrix (Other)
Collaborators: Banner University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16NE-GSAM-6364
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Hyperbilirubinemia
MeSH Terms: conditions — Hyperbilirubinemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Gestational Age 23 0/7 - 28 6/7 weeks
  Interventions: Diagnostic Test: TcB Measurement
- Group B: Gestational Age 29 0/7 weeks - 34 6/7 weeks
  Interventions: Diagnostic Test: TcB Measurement

INTERVENTIONS:
Diagnostic Test: TcB Measurement — TcB measurements will be obtained within approximately 30 minutes of the TSB being drawn before initiation of phototherapy, approximately 24 hours after the initiation of phototherapy and approximately 24 hours after completion of phototherapy. The TcB measurement will involve lightly pushing three times at each site which will yield an average transcutaneous bilirubin value. This will be calculated for the interscapular, buttock and sternal automatically by the bilirubinometer. While on phototherapy a measurement of the diapered, non-exposed buttock area will be obtained at approximately 24 hours to coincide with the standard of care serum bilirubin measurement.

SUMMARY:
The most common and widely accepted method of monitoring bilirubin levels in neonates is the use of the laboratory analyzation of serum blood levels. Unfortunately this method is invasive, painful, and can progressively lead to increased blood loss in the neonate. It also requires the use of additional time and resources to coordinate sending the sample to the laboratory and processing the specimen in the lab. There exists a different option for obtaining bilirubin levels in neonates which is the transcutaneous bilirubinometer. This device detects bilirubin levels at the bedside and has been validated for use in infants born at > 35 weeks gestation. There are a limited number of studies evaluating its use in premature infants.

Our aim is to assess the diagnostic accuracy and efficacy of transcutaneous bilirubinometry (TcB) of the Dräger JM-103 by comparing (TcB) readings to total serum bilirubin (TSB) results in neonates born at 23 0/7-34 6/7 weeks gestation.

DETAILED DESCRIPTION:
Design and Project Type In order to allow for appropriate data collection and comparison of TSB versus TcB measurements, this will be a prospective cohort study design. The expected duration will be 2 years. An interim analysis will occur approximately every six months.

Description of Intervention TcB measurements will be obtained within approximately 30 minutes of the TSB being drawn before initiation of phototherapy, approximately 24 hours after the initiation of phototherapy and approximately 24 hours after completion of phototherapy. The TcB measurement will involve lightly pushing three times at each site which will yield an average transcutaneous bilirubin value. This will be calculated for the interscapular, buttock and sternal automatically by the bilirubinometer. While on phototherapy a measurement of the diapered, non-exposed buttock area will be obtained at approximately 24 hours to coincide with the standard of care serum bilirubin measurement.

Instruments The JM-103 is the bilirubinometer that will be utilized in obtaining TcB measurements for this project. This meter is currently used on an as-needed basis within the unit for late preterm or term infants.

Data Collection Basic demographic data such as gestational age, ethnicity and gender will be collected. Relevant laboratory data such as blood type of mom and infant, and Coomb's test results will be collected. In addition, enteral and intravenous nutrition data will be collected including the type and volume of feeds at the same time the TcB is obtained. The results, date, time and location of the TSB and TcB will be collected for analysis.

TcB measurements will be obtained on those infants that are already ordered to have a blood draw for a serum bilirubin level. In the event the enrolled neonate does not require phototherapy during their hospitalization, the initial baseline TSB and TcB measurements will be collected and analyzed. Data will be collected during the first week of life. In the event that a neonate requires a second course of phototherapy and this is initiated during the first week of life, TcB and TSB measurements will be collected through the completion of phototherapy at 24 hours post treatment. If the enrolled neonate does not require phototherapy during their hospitalization, the initial baseline TSB and TcB measurements will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates with gestational age at delivery of 23 0/7 to 34 6/7 weeks

Exclusion Criteria:

* Neonates requiring blood exchange transfusion
* Lethal congenital anomalies
* Hydrops fetalis
* Infants who have received an intrauterine transfusion
* Investigator discretion as to other factors which might impact the study

Ages: 23 Weeks to 34 Weeks | Sex: All
Age Groups: Child
Study Population: Infants meeting gestational age criteria specified (23 0/7 up to 34 6/7 weeks gestation) without lethal congenital anomalies or hyperbilirubinemia requiring an exchange transfusion will be recruited for enrollment in this study. The enrolled babies will be divided into two groups based on gestational age as follows: Group A 23 0/7 - 28 6/7 weeks, and Group B 29 0/7 weeks - 34 6/7 weeks. A minimum of 60 infants will be enrolled into each group. As more subjects are likely to be eligible to be enrolled during the anticipated two year duration of the study, up to a maximum of 200 may be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
validity of transcutaneous bilirubin measurements | 2 years
  evaluate the validity of transcutaneous bilirubin measurements in premature infants born at 23 0/7- 28 6/7 weeks and 29 0/7 - 34 6/7 weeks gestation as compared to serum bilirubin measurements taken prior to, during and after phototherapy

SECONDARY OUTCOMES:
treatment with phototherapy | 2 years
  To compare transcutaneous bilirubin measurements obtained at different sites prior to and after treatment with phototherapy.
cost savings | 2 years
  To evaluate the cost savings of using the TcB meter measurements in place of the serum transcutaneous bilirubin

CONTACTS AND LOCATIONS:
Overall Officials: Suma Rao, MD, Principal Investigator — Pediatrix
Locations (1):
- Banner - University Medical Center Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Afanetti M, Eleni Dit Trolli S, Yousef N, Jrad I, Mokhtari M. Transcutaneous bilirubinometry is not influenced by term or skin color in neonates. Early Hum Dev. 2014 Aug;90(8):417-20. doi: 10.1016/j.earlhumdev.2014.05.009. Epub 2014 Jun 11. PMID 24951079
- [Background] Badiee Z, Mohammadizadeh M, Shamee M. Diagnostic usefulness of transcutaneous bilirubinometry in very preterm newborns. Int J Prev Med. 2012 Apr;3(4):262-5. PMID 22624082
- [Background] Grabenhenrich J, Grabenhenrich L, Buhrer C, Berns M. Transcutaneous bilirubin after phototherapy in term and preterm infants. Pediatrics. 2014 Nov;134(5):e1324-9. doi: 10.1542/peds.2014-1677. Epub 2014 Oct 20. PMID 25332501
- [Background] Karen T, Bucher HU, Fauchere JC. Comparison of a new transcutaneous bilirubinometer (Bilimed) with serum bilirubin measurements in preterm and full-term infants. BMC Pediatr. 2009 Nov 12;9:70. doi: 10.1186/1471-2431-9-70. PMID 19909530
- [Background] Maisels MJ, Bhutani VK, Bogen D, Newman TB, Stark AR, Watchko JF. Hyperbilirubinemia in the newborn infant > or =35 weeks' gestation: an update with clarifications. Pediatrics. 2009 Oct;124(4):1193-8. doi: 10.1542/peds.2009-0329. Epub 2009 Sep 28. No abstract available. PMID 19786452
- [Background] Nagar G, Vandermeer B, Campbell S, Kumar M. Reliability of transcutaneous bilirubin devices in preterm infants: a systematic review. Pediatrics. 2013 Nov;132(5):871-81. doi: 10.1542/peds.2013-1713. Epub 2013 Oct 14. PMID 24127472
- [Background] Rylance S, Yan J, Molyneux E. Can transcutaneous bilirubinometry safely guide phototherapy treatment of neonatal jaundice in Malawi? Paediatr Int Child Health. 2014 May;34(2):101-7. doi: 10.1179/2046905513Y.0000000050. Epub 2013 Dec 6. PMID 24090969
- [Background] Taylor JA, Burgos AE, Flaherman V, Chung EK, Simpson EA, Goyal NK, Von Kohorn I, Dhepyasuwan N; Better Outcomes through Research for Newborns Network. Discrepancies between transcutaneous and serum bilirubin measurements. Pediatrics. 2015 Feb;135(2):224-31. doi: 10.1542/peds.2014-1919. Epub 2015 Jan 19. PMID 25601981
- [Background] Varvarigou A, Fouzas S, Skylogianni E, Mantagou L, Bougioukou D, Mantagos S. Transcutaneous bilirubin nomogram for prediction of significant neonatal hyperbilirubinemia. Pediatrics. 2009 Oct;124(4):1052-9. doi: 10.1542/peds.2008-2322. Epub 2009 Sep 28. PMID 19786443